CLINICAL TRIAL: NCT01988142
Title: The Effect of Continuous Passive Motion Training on Neuromuscular Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Associate Professor, Chang Gung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 95-0973B
Record Dates: First submitted 2013-11-07; First posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Spinal Cord Injury(SCI)
Keywords: Spinal Cord Injury; Passive motion; Fatigue index; Hypertonia
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Hypertonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SCI (Experimental)
  Interventions: Procedure: Ankle continuous passive motion machine.

INTERVENTIONS:
Procedure: Ankle continuous passive motion machine. — A rehabilitation program of machine driven passive stretch.

SUMMARY:
After spinal cord injury (SCI), the muscular property altered due to the immobilization adaptation. The purpose of this study was to investigate the effect of remobilization with continuous passive exercise on the adapted paralyzed muscle properties after SCI.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic spinal cord injury

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Muscle tone tests | Baseline, 1, 2,3, and 4 months.
  Measure of changes in Hypertonia measured by Modified Ashworth Scale (MAS) and Patient Reported Impact of Spasticity Measure (PPSIM).
Fatigue index of muscle | Baseline, 1, 2,3, and 4 months.
  Measure of changes in Fatigue index of soleus and tibialis anterior (TA) muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan